CLINICAL TRIAL: NCT07299344
Title: Un Modello di Presa in Carico Continua Del Paziente Fragile
Brief Title: A Model for Continuous Care of Fragile Patients
Acronym: AFTER
Status: Not yet recruiting | Type: Observational
Sponsor: Azienda Sanitaria Locale CN2 Alba-Bra (Other)
Collaborators: Casa di Cura La Residenza di Rodello (CN, Italy) (Unknown)
Responsible Party: Sponsor
Other Study IDs: AFTER
Record Dates: First submitted 2025-11-28; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Neurological Disorders; Orthopedic Disorders; Functional Decline; Fragile and More Vulnerable
Keywords: Functional Monitoring; Functional Decline; Medically Fragile Patients; Neurological Disorders; Orthopedic Conditions; Rehabilitation; Proactive Care Model; Continuous Patient Management; Rehabilitation Setting; Early Detection of Functional Changes; telemedicine
MeSH Terms: conditions — Nervous System Diseases; Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Medically Fragile Patients with Neurological or Orthopedic Conditions: This cohort includes medically fragile adult patients with mild-to-moderate neurological or orthopedic conditions who are able to ambulate independently with or without assistive devices. Eligible neurological conditions include mild-to-moderate stroke (mRS ≤ 3), Multiple Sclerosis (EDSS ≤ 6.5), Parkinson's disease or parkinsonisms, and neuromuscular diseases. Eligible orthopedic conditions include femur, pelvis, or humerus fractures. Participants must have adequate cognitive function (MMSE ≥ 24) and the presence of a cognitively capable caregiver.
  Interventions: Other: Telemedicine-Based Functional Monitoring

INTERVENTIONS:
Other: Telemedicine-Based Functional Monitoring — This intervention provides structured functional monitoring of medically fragile patients with neurological and/or orthopedic conditions using telemedicine. Patients undergo MMSE, Rankin Scale, Barthel Index, TUG, GPCog, and SF-36 assessments at discharge and during follow-up at 3, 6, and 12 months. Patient and caregiver satisfaction with remote monitoring is also evaluated. All remote assessments are performed via the TESI eViSus BioCare® system on mobile devices, allowing early detection of functional decline and supporting proactive patient management.
  Other Names: Remote Functional Assessment Protocol; Telemedicine Follow-Up Monitoring

SUMMARY:
This observational study aims to monitor functional status and identify potential declines in the functioning of medically fragile patients with neurological and/or orthopedic conditions, representing an added value for ensuring appropriate patient management. This approach improves system efficiency and supports a proactive strategy that promotes the appropriate use of resources.

DETAILED DESCRIPTION:
This is a prospective, observational, non-profit study.

Primary Objective:

To compare functional and cognitive test results at discharge from "La Residenza" rehabilitation center (Rodello - CN- Italy) with remote assessments at patients' homes, demonstrating that Timed Up and Go (TUG) and GPCog tests, validated in-person, can be reliably administered via telemedicine.

Secondary Objectives:

To monitor motor and cognitive function remotely at 3, 6, and 12 months after discharge, assessing clinical course and disease progression, and evaluating patient condition as stable, improved, or deteriorated.

Study Timeline and Sample Size:

Recruitment is expected from September 2025 to March 2026, with last follow-up in March 2027 and an additional 6 months for data analysis and publication. A total of 100 patients (50 orthopedic, 50 neurological) will be enrolled, accounting for a 25% expected loss, based on power calculations for paired t-tests comparing in-person and remote assessments.

ELIGIBILITY:
Inclusion criteria:

* Adult medically fragile patients with one of the following neurological conditions: mild-to-moderate stroke (Rankin ≤ 3), Multiple Sclerosis (EDSS ≤ 6.5), Parkinson's disease or parkinsonisms, neuromuscular diseases; or orthopedic conditions: femur, pelvis, or humerus fracture.
* Able to walk independently, with or without assistive devices.
* Adequate cognitive function (MMSE ≥ 24).
* Patient or caregiver owns and can use a mobile device with internet/data connection.
* Presence of a cognitively capable, cooperative caregiver willing to participate in the study.

Exclusion criteria:

* Patients with severe neurological or orthopedic conditions who cannot walk independently, even with assistive devices.
* Patients with moderate or severe cognitive impairment (MMSE < 24).
* Patients with Barthel Index > 60.
* Patients or caregivers unable to use a mobile device or without internet/data connection.
* Patients without a cooperative, cognitively capable caregiver.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Medically fragile patients with various neurological or orthopedic conditions will be recruited from Casa di Cura "La Residenza" in Rodello (CN - Italy) for intensive rehabilitation. Patients will come from the Neurology and Orthopedics Units of Michele e Pietro Ferrero Hospital in Verduno (CN - Italy) - ASL CN2 .
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Concordance Between In-Person and Telemedicine Assessments of Functional and Cognitive Performance | 5-10 days after discharge
  Percentage of patients for whom the Timed Up and Go (TUG) test differs by less than 3.5 seconds and the GPCog test differs by less than 3 points between in-person and telemedicine assessments.

SECONDARY OUTCOMES:
Timed Up and Go (TUG) Test Performance | 3, 6, and 12 months after discharge
  The Timed Up and Go (TUG) test assesses functional mobility by measuring the time it takes (in seconds) for a participant to stand up from a chair, walk 3 meters, turn, walk back, and sit down. Lower times indicate better functional mobility.
  Unit of Measure: Seconds (s)
General Practitioner Assessment of Cognition (GPCog) Score | 3, 6, and 12 months after discharge
  General Practitioner Assessment of Cognition (GPCog), total score range 0-9. Higher scores indicate better cognitive functioning.
  Unit of Measure: Score on a scale (0-9)
Modified Rankin Scale (mRS) | Baseline and 12 months after discharge
  Modified Rankin Scale score assessing global disability. Range 0-6, where 0 = no symptoms and 6 = death. Higher scores indicate worse disability.
  Unit of Measure: Score on a scale (0-6)
Barthel Index for Activities of Daily Living | Baseline and 12 months after discharge
  Barthel Index score assessing independence in activities of daily living. Range 0-100. Higher scores indicate greater independence.
  Unit of Measure: Score on a scale (0-100)
SF-36 Composite Scores (Physical and Mental Component Summaries) | At discharge and 12 months after discharge
  Short Form-36 (SF-36) Health Survey assessing quality of life across multiple domains. Scores range 0-100 for each domain. Higher scores indicate better perceived health status.
  Unit of Measure: Score on a scale (0-100)
Patient Satisfaction With Remote Monitoring | 3, 6, and 12 months after discharge
  Patient satisfaction assessed using a validated satisfaction questionnaire (e.g., Likert scale 1-5). Higher scores indicate greater satisfaction.
  Unit of Measure: Score on a Likert scale (1-5)
Caregiver Satisfaction With Remote Monitoring | 3, 6, and 12 months after discharge
  Caregiver satisfaction assessed using a validated satisfaction questionnaire (e.g., Likert scale 1-5). Higher scores indicate greater satisfaction.
  Unit of Measure: Score on a Likert scale (1-5)

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Sanitaria Locale CN2 Alba-Bra, Ospedale Michele e Pietro Ferrero, Verduno, CN, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Feeney J, Savva GM, O'Regan C, King-Kallimanis B, Cronin H, Kenny RA. Measurement Error, Reliability, and Minimum Detectable Change in the Mini-Mental State Examination, Montreal Cognitive Assessment, and Color Trails Test among Community Living Middle-Aged and Older Adults. J Alzheimers Dis. 2016 May 31;53(3):1107-14. doi: 10.3233/JAD-160248. PMID 27258421
- [Background] Giavarina D. Understanding Bland Altman analysis. Biochem Med (Zagreb). 2015 Jun 5;25(2):141-51. doi: 10.11613/BM.2015.015. eCollection 2015. PMID 26110027
- [Background] Viglino G, Neri L, Barbieri S, Tortone C. Peritoneal dialysis training performed remotely: results and comparison with Home Training. Clin Exp Nephrol. 2023 Jan;27(1):72-78. doi: 10.1007/s10157-022-02276-z. Epub 2022 Sep 21. PMID 36129554
- [Background] Brodaty H, Pond D, Kemp NM, Luscombe G, Harding L, Berman K, Huppert FA. The GPCOG: a new screening test for dementia designed for general practice. J Am Geriatr Soc. 2002 Mar;50(3):530-4. doi: 10.1046/j.1532-5415.2002.50122.x. PMID 11943052
- [Background] van Dyck CH, Swanson CJ, Aisen P, Bateman RJ, Chen C, Gee M, Kanekiyo M, Li D, Reyderman L, Cohen S, Froelich L, Katayama S, Sabbagh M, Vellas B, Watson D, Dhadda S, Irizarry M, Kramer LD, Iwatsubo T. Lecanemab in Early Alzheimer's Disease. N Engl J Med. 2023 Jan 5;388(1):9-21. doi: 10.1056/NEJMoa2212948. Epub 2022 Nov 29. PMID 36449413
- [Background] de Joode SGCJ, Kalmet PHS, Fiddelers AAA, Poeze M, Blokhuis TJ. Long-term functional outcome after a low-energy hip fracture in elderly patients. J Orthop Traumatol. 2019 Apr 11;20(1):20. doi: 10.1186/s10195-019-0529-z. PMID 30976999